CLINICAL TRIAL: NCT04587284
Title: Economic Evaluation of Robot-assisted Laparoscopic Radical Prostatectomy vs Conventional Laparoscopic Radical Prostatectomy and Open Retropubic Radical Prostatectomy in Prostate Cancer: a Real-life Study Based on the French National Healthcare Data System (SNDS)
Acronym: ECOREPAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux PharmacoEpi (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/72
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with robot-assisted laparoscopic radical prostatectomy
- Patients with open retropubic radical prostatectomy
- Patients with laparoscopic radical prostatectomy

SUMMARY:
This study aims to assess the cost-effectiveness ratio and the clinical benefit (survival, disease recurrence, functional results) of the robot-assisted laparoscopic radical prostatectomy compared with other procedures using real-life data from SNDS. The population of patients who benefited from robot-assisted surgery will be identified in the SNDS through a practices survey, allowing the identification of centres fully converted to robotics.

DETAILED DESCRIPTION:
Over the last 15 years, robot-assisted laparoscopic radical prostatectomy surgery has seen a considerable rise in France. To date, it represents the most common surgical technique for radical prostatectomies, compared with standard procedure such as open retropubic radical prostatectomy or laparoscopic radical prostatectomy (8000 procedures/year, 40% of surgeries). In 2016, the French Health Authority (HAS) published a report on the robot-assisted laparoscopic radical prostatectomy practice that highlighted the small amount of available convincing data to provide evidence for a significant clinical benefit. There were no published data on overall or progression-free survival compared with other surgical procedures, with an important organizational and financial impact for healthcare institutions and patients. The question of the clinical benefit and the cost-effectiveness ratio of this surgical procedure is still relevant taking into account that randomized studies are difficult to carry out and that results of prospective registers will be available in many years. In this context, the use of the French National Claims Database (SNDS) appears to be the best short-term and reduced-cost solution to identify patients who benefited from the three surgical procedures since the rise of robotics. It would provide real-life data to national institutions in order to conclude on the opportunity to set a specific hospital tariff for the robot-assisted laparoscopic radical prostatectomy. This study aims to assess the cost-effectiveness ratio and the clinical benefit (survival, disease recurrence, functional results) of the robot-assisted laparoscopic radical prostatectomy compared with other procedures using real-life data from SNDS. The population of patients who benefited from robot-assisted surgery will be identified in the SNDS through a practices survey, allowing the identification of centres fully converted to robotics.

ELIGIBILITY:
Inclusion Criteria:

Total retro-pubic prostatectomy (PTRP) identified in the SNDS by the standard, Classification of Medical Acts "JGFA006" act

* Laparoscopic total prostatectomy (PTL) identified in the SNDS by the CCAM "JGFC001" act and the health and social establishment files number of centers not equipped with a surgical robot
* Robot-assisted total prostatectomy (PTRA) identified in the SNDS by the CCAM "JGFC001" act and the health and social establishment files number of centers equipped with a surgical robot for more than 12 months and having a rate of use of this technique for more than 95% minimally invasive prostatectomies. The number of PTRA will be identified by a survey in each center and the manufacturer's data as explained above

Patient who has not received previous treatment for this cancer by hormone therapy, radiotherapy, brachytherapy or HiFU (treatments sought in the SNDS prior to surgery by the prescription of pharmaceutical specialties or the presence of CCAM procedures)

Exclusion Criteria:

* Patient operated for laparoscopic radical prostatectomy or robot-assisted laparoscopic radical prostatectomy in a center equipped with a surgical robot but with a rate of use of this technique less than 95% (centers offering different minimally invasive approaches that do not allow to define if the intervention was performed in robotic surgery or in open surgery)
* Patient operated for a robot-assisted laparoscopic radical prostatectomy in a center having started a robotic activity for less than 12 months

Patient previously treated with another therapeutic modality for his prostate cancer (salvage prostatectomies after hormone therapy, radiotherapy, brachytherapy or HiFU)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups will be constituted according to surgical procedure: robot-assisted laparoscopic radical prostatectomy, open retropubic radical prostatectomy, and laparoscopic radical prostatectomy. All patients will be followed for at least 5 years and up to 8 years from the index date. Index date will be defined as the initial radical prostatectomy surgery performed between 2012-2015.
Sampling Method: Non-Probability Sample
Enrollment: 84667 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incremental cost / progression-free (without additional treatment) life-year saved 5 years after initial surgery | 5 years after initial surgery
  Progression-free survival requiring new treatment at 5 years will be calculated from :
  * Death within 5 years of surgery
  * Occurrence, over the period (5 years), of recurrences / progressions requiring additional treatment by radiotherapy and / or hormone therapy.
  A sensitivity analysis will be carried out after 1: 1 matching between subjects in each prostatectomy group.
  Estimation of the probability of event-free survival using the Kaplan-Meier estimator; Comparison of the risk of occurrence of each event between groups using a Cox proportional hazards model (after checking the underlying assumptions). The risk comparison will be measured using an hazard ratio, its 95% confidence interval and the p-value associated with the Wald test
  * without adjustment, from the overall population;
  * after adjustment for the propensity score, from the overall population;
  * from matched groups 1: 1.

SECONDARY OUTCOMES:
Incremental cost / life-year saved at 8 years. | 8 years after initial surgery
  Progression-free survival requiring new treatment at 5 years will be calculated from :
  * Death within 8 years of surgery
  * Occurrence, over the period (8 years), of recurrences / progressions requiring additional treatment by radiotherapy and / or hormone therapy.
  A sensitivity analysis will be carried out after 1: 1 matching between subjects in each prostatectomy group.
  Estimation of the probability of event-free survival using the Kaplan-Meier estimator; Comparison of the risk of occurrence of each event between groups using a Cox proportional hazards model (after checking the underlying assumptions). The risk comparison will be measured using an hazard ratio, its 95% confidence interval and the p-value associated with the Wald test
  * without adjustment, from the overall population;
  * after adjustment for the propensity score, from the overall population;
  * from matched groups 1: 1.

OTHER OUTCOMES:
Cost of robotic surgery. | 5 years after initial surgery;8 years after initial surgery
  None-adjusted estimation of cost-effectiveness ratios (95% confidence interval estimated by bootstrap) Net Monetary Benefit estimation of each surgical procedure (NMB = E x λ - C) with λ = differential cost-effectiveness threshold.
Urological hospitalizations within 90 days following the initial surgery. | 90 days following the initial surgery
  The initial hospital stay will be compared between the prostatectomy groups using standardized differences:
  * without adjustment, from the overall population;
  * after adjustment for the propensity score, from the overall population; from the matched groups 1: 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Talence, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robert G, Blin P, Bladou F, Jove J, Ouattara E, Rouyer M, Droz-Perroteau C, Piazza L, Preaubert N. Comparative effectiveness of robot-assisted vs. open prostatectomy: a real-life nationwide study. World J Urol. 2025 Jun 10;43(1):367. doi: 10.1007/s00345-025-05715-0. PMID 40493202